CLINICAL TRIAL: NCT06826261
Title: Home-based Transcranial Electrical Stimulation (tES) in Alzheimer's Disease
Brief Title: Digital Twins for Model-driven Non-invasive Electrical Brain Stimulation
Acronym: NEUROTWIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giacomo Koch, Prof, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101017716
Record Dates: First submitted 2025-01-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; tACS; brain stimulation; gamma
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHAM-tACS (Sham Comparator): The Sham condition will rely on the classical ramp up/ramp down protocol, which is characterized by 30 seconds of tACS stimulation at the beginning and end of the protocol to help with blinding. During the rest of the stimulation period (1h) no stimulation will be derivered.
  Interventions: Device: sham transcranial alternating current stimulation
- REAL-tACS (Experimental): The intervention will consist of daily model-optimized and individualized 40Hz-tACS delivered on the dorsolateral prefrontal and temporal cortex bilaterally. 40Hz-tACS will be applied daily for 1 hour, with a ramp up/down of 30 seconds.
  Interventions: Device: transcranial alternating current stimulation

INTERVENTIONS:
Device: transcranial alternating current stimulation — The intervention employs transcranial alternating current stimulation (tACS), a non-invasive brain stimulation technique designed to modulate neural oscillations in targeted brain regions. tACS operates by applying low-intensity, alternating electrical currents through electrodes placed on the scalp, synchronizing with the brain's natural frequency patterns. In this arm, a frequency of 40 Hz (gamma frequency) is used to enhance oscillatory activity related to cognitive functions often impaired in Alzheimer's disease (AD). The Neuroelectrics Starstim-home device will be used. This compact, portable device allows for easy use within the home setting, reducing the need for daily clinic visits. Designated caregivers will administer the one-hour tACS sessions under remote supervision via a digital monitoring portal, which tracks adherence, technical performance, and safety data in real time.
  Arms: REAL-tACS
Device: sham transcranial alternating current stimulation — The intervention employs transcranial alternating current stimulation (tACS), a non-invasive brain stimulation technique designed to modulate neural oscillations in targeted brain regions. tACS operates by applying low-intensity, alternating electrical currents through electrodes placed on the scalp, synchronizing with the brain's natural frequency patterns. In this arm, the stimulation will be delivered in 'sham' mode which is characterized by 30 seconds of tACS stimulation at the beginning and end of the protocol to help with blinding. During the rest of the stimulation period (1h) no stimulation will be delivered. The Neuroelectrics Starstim-home device will be used. This compact, portable device allows for easy use within the home setting, reducing the need for daily clinic visits. Designated caregivers will administer the sham tACS sessions under remote supervision via a digital monitoring portal, which tracks adherence, technical performance, and safety data in real time.
  Arms: SHAM-tACS

SUMMARY:
The purpose of this study is to obtain preliminary data in advance of a larger clinical trial designed to test whether repeated, daily sessions of at-home transcranial alternating current stimulation (tACS) can lead to a clinically significant improvement in patients with AD.

Given the potentially fragile patient population, the investigators propose a pilot study to test feasibility and safety (primary). In this pilot study 30 mild-to-moderate AD patients will be enrolled. The intervention will consist of daily model-optimized and individualized tES delivered for 8 weeks, 5 days per week (40 sessions). tACS will be applied daily for 1 hour and will be paired with extensive neuroimaging, neurophysiological and neuropsychological evaluation at several time points (pre and post treatment) to better characterize patients and their response to treatment. The physiological target of treatment will be to increase gamma activity in the pre-frontal cortex, as this has been associated with cognitive decline in AD, and prior tES work targeting PFC gamma oscillations has shown promising results.

The investigators hypothesize that active tACS treatment will result in a comparatively slower progression of cognitive decline and loss of gamma power as compared to sham treatment. To assess this, in this pilot study, a cross-over design will be used. Treatment will be multisession since prior tES work indicates a cumulative effect of each session with stronger therapeutic effects, in line with the underlying Hebbian mechanisms putatively involved in non-invasive brain stimulation.

DETAILED DESCRIPTION:
The NEUROTWIN project is grounded in the hypothesis that brain oscillations, particularly in the gamma band (40 Hz), play a central role in cognitive processes, and their disruption is associated with the cognitive decline seen in Alzheimer's disease (AD). Gamma oscillations are generated by excitatory-inhibitory neural circuits that include GABAergic interneurons, which are often impaired in patients with AD. This deficit is linked to reduced synchronization of gamma oscillations, which are essential for cognitive functions such as memory and attention.

Recent studies have shown that inducing gamma oscillations can reduce levels of amyloid-beta (Aβ) and phosphorylated tau (p-tau)-key pathological markers of AD-in animal models of the disease. These findings suggest that stimulating gamma oscillations through non-invasive methods may have a positive impact on specific brain functions affected by AD. Transcranial electrical stimulation (tES), including transcranial alternating current stimulation (tACS), can modulate these gamma oscillations in a safe, non-invasive manner.

The rationale for targeting gamma oscillations with tACS in Alzheimer's therapy is supported by:

* Preclinical and clinical evidence: Studies in murine AD models have demonstrated a significant reduction in amyloid plaques and p-tau levels in mice exposed to gamma stimulation (40 Hz), along with cognitive improvements.
* Previous clinical experiments: The use of 40 Hz tACS has enhanced episodic memory and cerebral perfusion in small cohorts of human patients with AD. These preliminary results indicate that gamma stimulation may represent a promising therapeutic approach for modulating cognitive function in AD patients.
* Impact of neural dysfunction in AD: Dysfunction in neural circuits, especially involving inhibitory interneuron control, can lead to an excitatory-inhibitory imbalance, resulting in cognitive impairments. Stimulating gamma oscillations may improve the function of altered neural circuits, contributing to cognitive stabilization.

However, a significant constraint of many Non-invasive brain stimulation protocols is their reliance on multiple sessions to achieve enduring effects. These sessions are typically conducted in clinical settings, necessitating patient travel. This obstacle hampers the delivery of extended interventions, particularly for individuals with neurodegenerative conditions. We thus adopt a home-based approach using tACS because of its ability to entrain gamma oscillations, commonly impaired in AD, and its low cost and potential for home-based application. in particular, the Starstim-home device has been developed for home use with remote supervision, making gamma stimulation accessible and scalable for patients. A home-based protocol allows for a higher treatment frequency (5 times a week for 8 weeks per arm), reducing costs and increasing convenience for patients and caregivers.

In this study, participants will use the Starstim-home device for one-hour tACS sessions (real or sham), targeting the fronto-temporal cortex. These electrode positions were obtained from a group montage optimization using the Stimweaver algorithm performed on a database of biophysical head models of patients with AD, i.e. volume conductor models built from structural head T1w-MRIs that model the passive electrical properties of the primary head tissues.

The device will be configured to administer personalized and model-optimized gamma-frequency tES, always assuming a 180° phase-shift between the currents in the electrodes in the opposite hemispheres. This is done using a linear model that predicts the currents based on morphometric characteristics of the patient's scalp, namely the head perimeter along axial, sagittal, and coronal planes. The current intensity will be ramped up over the first 30 seconds, then sustained at the stimulation intensity for 60 minutes, then ramped down over the final 30 seconds for the Real condition. The Sham condition will rely on the classical 30-second ramp-up/ramp-down protocol.

The subject will receive a pre-configured Starstim Home Kit, including the device, tablet, all needed supplies, and training materials. The Starstim Home Kit tablet contains a sequence of simplified instructions and step-by-step touchscreen prompts for the participant/administrator to follow. This process has been designed to be easy to use, even for individuals who are not computer savvy.

The first two daily visits will be performed at the memory clinic. During the first daily visit, the study staff will lead a training session while the home-based administrator observes. The study staff will review the step-by-step process, the accompanying training manual, and the photos depicting each step. During the second daily visit, the administrator will then practice setting up the tES session on the participant with oversight and coaching from the study staff. The administrator will also be trained to take care of the devices. Then, caregivers or designated administrators will oversee the sessions at home, ensuring device use and protocol adherence under remote supervision by clinical staff.

In this randomized, double-blind, sham-controlled, crossover pilot study, the participants will receive both active and sham tES conditions, each lasting 8 weeks, with a washout period of two months in between. tES sessions will be held daily, 5 days a week, for a total of 40 sessions per condition. Neuroimaging, neurophysiological, and cognitive assessments will occur at multiple points before, after, and in a follow-up period of two months for each treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50 and 85.
* Clinical Dementia Rating score (CDR) of 0.5-1.
* Mini-Mental State Examination (MMSE) score of 18-26.
* treated with acetylcholinesterase inhibitor for at least one month.
* evidence of low β-amyloid and/or elevated phosphorylated Tau protein as detected by lumbar puncture for cerebrospinal fluid biomarkers analysis for diagnostic purposes or PET.
* have a Caregiver
* have access to wireless internet (wifi) connection in the location where study treatments will be applied

Exclusion Criteria:

* significant neurodegenerative disorder of the central nervous system other than AD.
* significant intracranial focal or vascular pathology verified by an MRI scan.
* history of seizures (except febrile seizures in childhood).
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM IV-TR) criteria met for any of the following (within the specified period): Major depressive disorder (current), Schizophrenia (lifetime), Other psychotic disorders, bipolar disorder, or substance (including alcohol) related disorders (within the past 5 years).
* contraindications to MRI (this includes metal implants in the head, pacemaker, cochlear implants, or any other non-removable items if they are contraindications to MR imaging).
* treatment currently or within 3 months before Baseline with any of the following medications: typical and atypical antipsychotics (i.e., Clozapine, Olanzapine); antiepileptics drugs (i.e., Carbamazepine, Primidone, Pregabalin, Gabapentin).
* skin lesions on the scalp at the proposed electrode sites.
* previous surgeries opening the skull leaving skull defects capable of allowing the insertion of a cylinder with a radius greater or equal to 5 mm.
* any condition that makes the study subject, in the opinion of the investigator, unsuitable for the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events and missed stimulation session | From date of randomization until the date of last documented progression, assessed up to 8 months
  The investigators will collect data about electrode impedance, tACS progression, and session interruptions or terminations, whether voluntary or due to technical issues. These metrics, including the number of missed sessions, will aid in the assessment of feasibility. At the same time, any adverse events will be documented and used as the primary safety endpoint.
Measurement of change from baseline in the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) 14 immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) 14 is a standardized neuropsychological assessment used to measure the severity of symptoms of Alzheimer's Disease in different domains. The tasks assess the domains of language, praxis, memory, attention, visuospatial and executive function. The tasks include: word recall task, naming objects and fingers, commands, constructional praxis, ideational praxis, orientation, word recognition task, comprehension of spoken language, word finding difficulty, remembering test instructions, executive function, and number cancellation. The score range is from 0 to 70 with a lower score indicating more severe functional impairment.

SECONDARY OUTCOMES:
Measurement of change from baseline in the Clinical Dementia Rating scale (C.D.R.) sum of boxes immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The Clinical Dementia Rating scale (C.D.R.) sum of boxes is used to characterize six domains of cognitive and functional performance applicable to Alzheimer's disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. The score range is from 0 to 18 with the higher score meaning greater disease severity.
Measurement of change from baseline in the AD Cooperative Study - Activities of Daily Living (ADCS-ADL) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The AD Cooperative Study - Activities of Daily Living (ADCS-ADL) includes 23 items that were derived from a larger set of items describing the performance of activities of daily living. The score range is from 0 to 78 with a lower score indicating more severe functional impairment.
Measurement of change from baseline in the Mini-Mental State Examination (MMSE) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The Mini-Mental State Examination (MMSE) is a brief, widely used valid, and reliable assessment of cognitive impairment. This 30-point questionnaire is used to screen and estimate the severity of cognitive impairment in addition to being used to follow the course of cognitive change over time. The test assesses orientation, attention and calculation, recall, language, repetition, and ability to follow complex commands. The score range is from 0 to 30, with lower score meaning greater cognitive impairment.
Measurement of change from baseline in the Frontal Assessment Battery (F.A.B.) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The Frontal Assessment Battery (F.A.B.) is a brief battery of six neuropsychological tasks designed to assess frontal lobe function at the bedside. The six FAB tasks explore cognitive and behavioral domains that are thought to be under the control of the frontal lobes, most notably conceptualization, and abstract reasoning, lexical verbal fluency and mental flexibility, motor programming and executive control of action, self-regulation, and resistance to interference, inhibitory control, and environmental autonomy. The range score is from 0 to 18 with the higher score meaning less frontal cognitive impairment.
Measurement of change from baseline in the Neuropsychiatric Inventory (NPI) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The Neuropsychiatric Inventory assesses behavioral disturbances in dementia. The NPI is a reliable and valid test measuring the following behavioral areas: delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor behavior, night time behaviors, and eating disorders. The score range is from 0 to 144 with the higher score meaning more severe behavioural disturbances.
Measurement of change from baseline in the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form is a 16-item, self-report questionnaire that evaluates quality of life and satisfaction in several domains. The first 14 items assess satisfaction with (1) physical health, (2) mood, (3) work, (4) household activities, (5) social relationships, (6) family relationships, (7) leisure activities, (8) daily functioning, (9) sexual life, (10) economic status, (11) living/housing situation, (12) ability to get around physically, (13) vision, and (14) overall well-being. The last two items measure medications, and overall satisfaction and contentment. The items are scored on a 5-point Likert scale from 1 (not at all or never) to 5 (frequently or all the time), with higher scores indicating better enjoyment and satisfaction with life. The total score of the questionnaire is the sum of these 14 items ranging from 14 to 70. Higher scores mean better enjoyment and satisfaction with life.
Measurement of change from baseline in the Apathy Motivation Index immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The apathy motivation index is a 18-item self-report questionnaire that assesses apathy in terms of Behavioral Activation (tendency to self-initiate goal-directed behavior), Social Motivation (level of engagement in social interactions) and Emotional Sensitivity (affective responses) using a 5-point Likert scale. Item scores are averaged to yield scores for subscales and a total score with higher scores indicating greater apathy (range 0-4).

OTHER OUTCOMES:
Measurement of change from baseline in the Resting-state EEG activity in specific frequency band of relevance for AD immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  Resting state EEG and artifact recordings will be obtained by using 64 channels TMS-compatible EEG equipment (BrainAmp 32MRplus, BrainProducts GmbH, Munich, Germany) with the eyes open for five minutes.
Measurement of change from baseline in the short afferent inhibition (SAI) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  This measure reflects the central cholinergic activity controlled by inhibitory circuits.
Measurement of change from baseline in the Repetitive TMS indexing long term potentiation (LTP) immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
Measurement of change from baseline in the transcranial evoked potentials (TEPs) and oscillatory activity over the fronto-temporal cortices immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  TMS-EEG protocol will be used to investigate changes in cortical reactivity, connectivity, and oscillatory evoked activity. A 64-channel TMS-compatible EEG equipment (BrainAmp 32MRplus, BrainProducts GmbH, Munich, Germany) will be used to collect data. A masking noise system will be used to reduce auditory evoked potential artifacts. The stimulation will take place over brain regions in the prefrontal and parietal lobes.
Measurement of change from baseline in the functional and structural connectivity immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  The MRI imaging will be conducted on a 3T Siemens Magnetom Prisma scanner with a 64-channel head-neck coil at the Neuroimaging department of IRCCS Santa Lucia Foundation (Rome, Italy). The subjects will be instructed to maintain their eyes open fixing a cross, not to focus their thoughts on any particular topic, and not to cross their arms or legs. The following sequences will be collected: Anatomical MRI, Diffusion MRI, Resting-state BOLD fMRI, and Resting-state ASL.
Measurement of change from baseline in the Blood biomarkers immediately after the intervention and at a two-month follow-up | From date of randomization until the date of last documented progression, assessed up to 8 months
  Blood biomarkers will be collected to detect plasmatic changes in amyloid beta, phosphorylated tau, and total tau, neurofilament light chain (NFL) (PG/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Bonni, PhD, Study Chair — I.R.C.C.S. Fondazione Santa Lucia; Martina Assogna, MD, Study Director — I.R.C.C.S. Fondazione Santa Lucia
Locations (1):
- Irccs Santa Lucia Foundation, Rome, ROME, Italy

IPD SHARING:
Plan to Share IPD: Yes
This study is part of the 'Horizon 2020' project and all data will be made publicly available in a digital database at the conclusion of the study.
Supporting Information: Study Protocol, ICF
Time Frame: 30/06/2025
Access Criteria: The IPD supporting information will be made available upon request and accessed using a password.

REFERENCES:
- [Background] Dhaynaut M, Sprugnoli G, Cappon D, Macone J, Sanchez JS, Normandin MD, Guehl NJ, Koch G, Paciorek R, Connor A, Press D, Johnson K, Pascual-Leone A, El Fakhri G, Santarnecchi E. Impact of 40 Hz Transcranial Alternating Current Stimulation on Cerebral Tau Burden in Patients with Alzheimer's Disease: A Case Series. J Alzheimers Dis. 2022;85(4):1667-1676. doi: 10.3233/JAD-215072. PMID 34958021
- [Background] Thickbroom GW. Transcranial magnetic stimulation and synaptic plasticity: experimental framework and human models. Exp Brain Res. 2007 Jul;180(4):583-93. doi: 10.1007/s00221-007-0991-3. Epub 2007 Jun 12. PMID 17562028
- [Background] Tadini L, El-Nazer R, Brunoni AR, Williams J, Carvas M, Boggio P, Priori A, Pascual-Leone A, Fregni F. Cognitive, mood, and electroencephalographic effects of noninvasive cortical stimulation with weak electrical currents. J ECT. 2011 Jun;27(2):134-40. doi: 10.1097/YCT.0b013e3181e631a8. PMID 20938352
- [Background] Sprugnoli G, Munsch F, Cappon D, Paciorek R, Macone J, Connor A, El Fakhri G, Salvador R, Ruffini G, Donohoe K, Shafi MM, Press D, Alsop DC, Pascual Leone A, Santarnecchi E. Impact of multisession 40Hz tACS on hippocampal perfusion in patients with Alzheimer's disease. Alzheimers Res Ther. 2021 Dec 20;13(1):203. doi: 10.1186/s13195-021-00922-4. PMID 34930421
- [Background] Ruffini G, Fox MD, Ripolles O, Miranda PC, Pascual-Leone A. Optimization of multifocal transcranial current stimulation for weighted cortical pattern targeting from realistic modeling of electric fields. Neuroimage. 2014 Apr 1;89:216-25. doi: 10.1016/j.neuroimage.2013.12.002. Epub 2013 Dec 15. PMID 24345389
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Palm U, Kumpf U, Behler N, Wulf L, Kirsch B, Worsching J, Keeser D, Hasan A, Padberg F. Home Use, Remotely Supervised, and Remotely Controlled Transcranial Direct Current Stimulation: A Systematic Review of the Available Evidence. Neuromodulation. 2018 Jun;21(4):323-333. doi: 10.1111/ner.12686. Epub 2017 Sep 15. PMID 28913915
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Mohs RC, Knopman D, Petersen RC, Ferris SH, Ernesto C, Grundman M, Sano M, Bieliauskas L, Geldmacher D, Clark C, Thal LJ. Development of cognitive instruments for use in clinical trials of antidementia drugs: additions to the Alzheimer's Disease Assessment Scale that broaden its scope. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S13-21. PMID 9236948
- [Background] Miranda PC, Mekonnen A, Salvador R, Ruffini G. The electric field in the cortex during transcranial current stimulation. Neuroimage. 2013 Apr 15;70:48-58. doi: 10.1016/j.neuroimage.2012.12.034. Epub 2012 Dec 27. PMID 23274187
- [Background] Magni E, Binetti G, Bianchetti A, Rozzini R, Trabucchi M. Mini-Mental State Examination: a normative study in Italian elderly population. Eur J Neurol. 1996 May;3(3):198-202. doi: 10.1111/j.1468-1331.1996.tb00423.x. PMID 21284770
- [Background] Koch G, Di Lorenzo F, Bonni S, Ponzo V, Caltagirone C, Martorana A. Impaired LTP- but not LTD-like cortical plasticity in Alzheimer's disease patients. J Alzheimers Dis. 2012;31(3):593-9. doi: 10.3233/JAD-2012-120532. PMID 22647254
- [Background] Galasko D, Schmitt F, Thomas R, Jin S, Bennett D; Alzheimer's Disease Cooperative Study. Detailed assessment of activities of daily living in moderate to severe Alzheimer's disease. J Int Neuropsychol Soc. 2005 Jul;11(4):446-53. doi: 10.1017/s1355617705050502. PMID 16209425
- [Background] Chiaravalloti A, Koch G, Toniolo S, Belli L, Lorenzo FD, Gaudenzi S, Schillaci O, Bozzali M, Sancesario G, Martorana A. Comparison between Early-Onset and Late-Onset Alzheimer's Disease Patients with Amnestic Presentation: CSF and (18)F-FDG PET Study. Dement Geriatr Cogn Dis Extra. 2016 Apr 5;6(1):108-19. doi: 10.1159/000441776. eCollection 2016 Jan-Apr. PMID 27195000
- [Background] Chiaravalloti A, Martorana A, Koch G, Toniolo S, di Biagio D, di Pietro B, Schillaci O. Functional correlates of t-Tau, p-Tau and Abeta(1)(-)(4)(2) amyloid cerebrospinal fluid levels in Alzheimer's disease: a (1)(8)F-FDG PET/CT study. Nucl Med Commun. 2015 May;36(5):461-8. doi: 10.1097/MNM.0000000000000272. PMID 25646706
- [Background] Charvet LE, Kasschau M, Datta A, Knotkova H, Stevens MC, Alonzo A, Loo C, Krull KR, Bikson M. Remotely-supervised transcranial direct current stimulation (tDCS) for clinical trials: guidelines for technology and protocols. Front Syst Neurosci. 2015 Mar 17;9:26. doi: 10.3389/fnsys.2015.00026. eCollection 2015. PMID 25852494
- [Background] Casula EP, Borghi I, Maiella M, Pellicciari MC, Bonni S, Mencarelli L, Assogna M, D'Acunto A, Di Lorenzo F, Spampinato DA, Santarnecchi E, Martorana A, Koch G. Regional Precuneus Cortical Hyperexcitability in Alzheimer's Disease Patients. Ann Neurol. 2023 Feb;93(2):371-383. doi: 10.1002/ana.26514. Epub 2022 Oct 18. PMID 36134540
- [Background] Casula EP, Pellicciari MC, Bonni S, Borghi I, Maiella M, Assogna M, Minei M, Motta C, D'Acunto A, Porrazzini F, Pezzopane V, Mencarelli L, Roncaioli A, Rocchi L, Spampinato DA, Caltagirone C, Santarnecchi E, Martorana A, Koch G. Decreased Frontal Gamma Activity in Alzheimer Disease Patients. Ann Neurol. 2022 Sep;92(3):464-475. doi: 10.1002/ana.26444. Epub 2022 Jul 7. PMID 35713198
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Andre S, Heinrich S, Kayser F, Menzler K, Kesselring J, Khader PH, Lefaucheur JP, Mylius V. At-home tDCS of the left dorsolateral prefrontal cortex improves visual short-term memory in mild vascular dementia. J Neurol Sci. 2016 Oct 15;369:185-190. doi: 10.1016/j.jns.2016.07.065. Epub 2016 Jul 30. PMID 27653887
- [Background] Koch G, Bonni S, Pellicciari MC, Casula EP, Mancini M, Esposito R, Ponzo V, Picazio S, Di Lorenzo F, Serra L, Motta C, Maiella M, Marra C, Cercignani M, Martorana A, Caltagirone C, Bozzali M. Transcranial magnetic stimulation of the precuneus enhances memory and neural activity in prodromal Alzheimer's disease. Neuroimage. 2018 Apr 1;169:302-311. doi: 10.1016/j.neuroimage.2017.12.048. Epub 2017 Dec 19. PMID 29277405
- [Background] Agarwal S, Pawlak N, Cucca A, Sharma K, Dobbs B, Shaw M, Charvet L, Biagioni M. Remotely-supervised transcranial direct current stimulation paired with cognitive training in Parkinson's disease: An open-label study. J Clin Neurosci. 2018 Nov;57:51-57. doi: 10.1016/j.jocn.2018.08.037. Epub 2018 Sep 5. PMID 30193898
- See also: Related Info — https://www.neurotwin.eu/